CLINICAL TRIAL: NCT07273227
Title: A Multicenter Randomized Controlled Trial of Echocardiography-Guided Atrial Septal Defect Closure Performed in a Mobile Surgical Unit
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Cheng Wang, Principal Investigator, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-2488
Record Dates: First submitted 2025-11-23; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: ASD - Atrial Septal Defect
Keywords: echocardiography-guided; percutaneous intervention; atrial septal defect; mobile surgical vehicle; mobile surgical unit
MeSH Terms: conditions — Heart Septal Defects, Atrial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Surgical Vehicle Echocardiography-guided ASD closure Group (Experimental): Patients undergo ultrasound-guided percutaneous atrial septal defect closure performed inside a mobile surgical vehicle.
  Interventions: Other: Mobile Surgical Vehicle Echocardiography-guided ASD closure Group
- Conventional Operating Room Echocardiography-guided ASD closure Group (Active Comparator): Patients undergo ultrasound-guided percutaneous atrial septal defect closure performed in a conventional operating room.
  Interventions: Other: Conventional Operating Room Echocardiography-guided ASD closure Group

INTERVENTIONS:
Other: Mobile Surgical Vehicle Echocardiography-guided ASD closure Group — Patients undergo ultrasound-guided percutaneous atrial septal defect closure performed inside a mobile surgical vehicle.
  Arms: Mobile Surgical Vehicle Echocardiography-guided ASD closure Group
Other: Conventional Operating Room Echocardiography-guided ASD closure Group — Patients undergo ultrasound-guided percutaneous atrial septal defect closure performed in a conventional operating room.
  Arms: Conventional Operating Room Echocardiography-guided ASD closure Group

SUMMARY:
Cardiovascular disease remains a major threat to global health, and structural heart disease which encompassing congenital heart defects, valvular disease, and cardiomyopathies constitutes a substantial proportion of its burden. Atrial septal defect (ASD) is among the most common congenital heart conditions, occurring in approximately 1.6 per 1,000 live births. Percutaneous closure of ASD has become the standard treatment due to its minimally invasive nature and proven efficacy. However, conventional closure procedures rely heavily on fluoroscopic guidance and iodinated contrast, which carry risks of radiation exposure, contrast-related harm, and limit applicability in specific patient groups. Moreover, such procedures must be performed in catheterization laboratories equipped with digital subtraction angiography systems.

To overcome these limitations, our team has spent over a decade developing a fully ultrasound-guided, radiation-free, contrast-free percutaneous intervention system-an original Chinese innovation that has pioneered "no incision, no fluoroscopy, and no general anesthesia" treatment for structural heart disease. This methodology has evolved into a comprehensive technical system and has been successfully applied to ASD, PFO, ventricular septal defect (VSD), patent ductus arteriosus (PDA), and several valvular disorders. It has been recognized by national clinical guidelines (2017), awarded the Chinese Medical Association First-Class Science and Technology Award (2022), and honored by the World Health Organization Innovation Award.

Building upon the unique advantages of ultrasound-only guidance, we further developed a Mobile Surgical Vehicle. This mobile surgical unit integrates ultrasound imaging, sterilization, monitoring, and anesthesia equipment, enabling true "hospital-free" procedures for underserved regions lacking large medical devices. Early applications in remote areas of Southwest China and Belt-and-Road countries have demonstrated promising safety and feasibility.

Nevertheless, high-quality clinical evidence evaluating this mobile platform for ASD closure is lacking. To address this gap, we propose a multicenter randomized controlled trial to demonstrate that mobile-platform ultrasound-guided closure is non-inferior to conventional in-hospital ultrasound-guided procedures. This study will also refine methodology, workflow, and safety protocols for mobile interventional therapy. Its findings will provide essential evidence supporting this original Chinese technology, expand its international impact, and enable broader access for patients in remote regions.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥8 years and able to undergo percutaneous intervention under local anesthesia.
* Diagnosed with secundum ASD with a defect diameter of ≥6 mm and ≤36 mm, accompanied by right-sided volume overload.
* Anatomical features suitable for transcatheter closure: the distance from the defect rim to the coronary sinus, superior vena cava, inferior vena cava, and pulmonary veins is ≥5 mm; and the distance to the mitral valves is ≥7 mm.

Exclusion Criteria:

* Presence of primum ASD or sinus venosus ASD.
* Infective endocarditis or intracardiac thrombus.
* ASD with right-to-left shunting.
* Concomitant intracardiac anomalies requiring simultaneous surgical repair.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-12-19 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
composite endpoint events | at 30 days after the procedure
  Composite endpoint events at 30 days after procedure, including failure of ultrasound-guided closure (conversion to fluoroscopy-guided intervention or open-heart surgery), residual shunt >2 mm, device embolization or migration, new-onset arrhythmia, bleeding, and infection.

SECONDARY OUTCOMES:
failure of ultrasound-guided closure (conversion to fluoroscopy-guided intervention or open-heart surgery) | immediately after the procedure
  failure of ultrasound-guided closure (conversion to fluoroscopy-guided intervention or open-heart surgery)
residual shunt >2 mm | at 30 days after the procedure
  residual shunt >2 mm under echocardiography
device embolization or migration | at 30 days after the procedure
  new device embolization or migration after procedure
new-onset arrhythmia | at 30 days after the procedure
  new-onset arrhythmia after procedure
bleeding | at 30 days after the procedure
  new bleeding after the procedure
infection | at 30 days after the procedure
  new infection after procedure
Composite endpoint events at 1 year | at 1 year after the procedure
  Composite endpoint events at 1 year after procedure, including failure of ultrasound-guided closure (conversion to fluoroscopy-guided intervention or open-heart surgery), residual shunt >2 mm, device embolization or migration, new-onset arrhythmia, bleeding, and infection.
length of postoperative hospital stay | at discharge (within 10 days after the procedure)
  length of postoperative hospital stay
hospitalization costs | at discharge (within 10 days after the procedure)
  hospitalization cost

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences, Fuwai Hospital, Beijing, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided